CLINICAL TRIAL: NCT01627665
Title: New Oral Anticoagulant Drugs Dabigatran Etexilate and Rivaroxaban: Influence of Genetic Factors in Healthy Volunteers
Brief Title: Pharmacogenomic Study on PKD/PKC of Dabigatran Etexilate and Rivaroxaban
Acronym: DRIVING
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: P081208
Record Dates: First submitted 2012-04-27; First posted 2012-06-26 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2011-03

CONDITIONS: Healthy Volunteers
Keywords: dabigatran; rivaroxaban; PKC; PKD; p-glycoprotein; polymorphism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- D->R->C+R (Active Comparator): sequence of treatment: Dabigatran after rivaroxaban after chlarythromycin in association with rivaroxaban
  Interventions: Drug: D->R->C+R
- D->R->C+D (Active Comparator): sequence of treatment: Dabigatran after rivaroxaban after chlarythromycin in association with Dabigatran
  Interventions: Drug: D->R->C+D
- R->D->C+D (Active Comparator): sequence of treatment: rivaroxaban after Dabigatran after chlarythromycin in association with Dabigatran
  Interventions: Drug: R->D->C+D
- R->D->C+R (Active Comparator): sequence of treatment: rivaroxaban after Dabigatran after chlarythromycin in association with rivaroxaban
  Interventions: Drug: R->D->C+R

INTERVENTIONS:
Drug: D->R->C+R — one oral dose DABIGATRAN 300 mg -> RIVAROXABAN 40 mg -> 1g/day CLARITHOMYCINE with RIVAROXABAN 40 mg
  Arms: D->R->C+R
Drug: D->R->C+D — one oral dose DABIGATRAN 300 mg -> RIVAROXABAN 40 mg -> 1g/day CLARITHOMYCINE with one oral dose DABIGATRAN 300 mg
  Arms: D->R->C+D
Drug: R->D->C+D — RIVAROXABAN 40 mg -> one oral dose DABIGATRAN 300 mg -> 1g/day CLARITHOMYCINE with one oral dose DABIGATRAN 300 mg
  Arms: R->D->C+D
Drug: R->D->C+R — RIVAROXABAN 40 mg -> one oral dose DABIGATRAN 300 mg -> 1g/day CLARITHOMYCINE with RIVAROXABAN 40 mg
  Arms: R->D->C+R

SUMMARY:
The study will address the impact of genetical variation of a protein involved in the intestinal absorption of two new anticoagulants : Dabigatran etexilate and Rivaroxaban.

DETAILED DESCRIPTION:
The study will address the impact of genetical variation of a protein involved in the intestinal absorption of two new anticoagulants : Dabigatran etexilate and Rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* Aged between 18-35 years inclusive
* Male
* Caucasian
* Body mass index (BMI) between 18 and 27 kg per m² inclusive.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2011-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
AUC of plasma concentrations of the drugs | over 24h after single oral dose

SECONDARY OUTCOMES:
PKD of the drugs | over 24h after single oral dose

CONTACTS AND LOCATIONS:
Overall Officials: Anne Blanchard, MD, Principal Investigator — CIC HEGP
Locations (1):
- CIC Hopital europeen george pompidou, Paris, Paris, France

REFERENCES:
- [Derived] Foulon-Pinto G, Jourdi G, Perrin J, Abdoul J, Paris G, Gouin-Thibault I, Curis E, Lecompte T, Siguret V. Study of thrombin generation with St Genesia to evaluate xaban pharmacodynamics: Analytical performances over 18 months. Int J Lab Hematol. 2021 Aug;43(4):821-830. doi: 10.1111/ijlh.13443. Epub 2020 Dec 28. PMID 33369212
- [Derived] Marques P, Courand PY, Gouin-Thibault I, Zhygalina V, Bergerot D, Salem JE, Funck-Brentano C, Loriot MA, Azizi M, Blanchard A. P-glycoprotein influences urinary excretion of aldosterone in healthy individuals. J Hypertens. 2019 Nov;37(11):2225-2231. doi: 10.1097/HJH.0000000000002150. PMID 31157746